CLINICAL TRIAL: NCT05849571
Title: Investigation of the Effect of Oral Care With Coconut Oil on the Degree of Oral Mucositis in Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Büşra Ekinci (Other)
Responsible Party: Sponsor-Investigator, Büşra Ekinci, Nurse, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-13022260-199-309276
Record Dates: First submitted 2023-02-04; First posted 2023-05-09 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Oral Mucositis
Keywords: oral mucositis; child; cancer; Oral care; Nursing; coconut oil
MeSH Terms: conditions — Stomatitis; Neoplasms | interventions — Coconut Oil

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control group (No Intervention): * Consent is obtained with an informed consent form.
  * Patient identification form is filled.
  * The patient's mouth is evaluated using the World Health Organization Mucositis Classification and the International Pediatric Mucositis Rating Scale (ChIMES) before receiving chemotherapy. According to the World Health Organization Mucositis Classification, the frequency of oral care is decided.
  * The patient's mouth is evaluated using the World Health Organization Mucositis Classification and the International Child Mucositis Evaluation Scale (ChIMES) on days 0, 7, and 14, and after each assessment, the frequency of oral care is determined and applied for 21 days. The final assessment is made on Day 21.
  * The care given according to the frequency of oral care determined according to the score obtained by the patient in the World Health Organization Mucositis Classification is recorded on the "Basic Oral Care Protocol Follow-up Chart".
- Experimental: Experimental Group (Experimental): Unlike the control group, the experimental group is rinsed with 5 ml of coconut 4 times a day.
  Interventions: Other: coconut oil

INTERVENTIONS:
Other: coconut oil — • The patient's mouth is evaluated using the World Health Organization Mucositis Classification and the International Child Mucositis Evaluation Scale (ChIMES) on days 0, 7, and 14, and after each assessment, the frequency of oral care is determined and applied for 21 days. The final assessment is made on Day 21.
  Arms: Experimental: Experimental Group

SUMMARY:
Oral mucositis is characterized by ulcerative and inflammatory changes in the oral mucosa and is frequently seen in pediatric oncology patients receiving chemotherapy. Oral mucositis negatively affects the child's daily life functions, nutrition and quality of life. Pain is the most commonly reported side effect in mucositis. Pain impairs patients' ability to chew, swallow and speak, leading to inadequate fluid/nutrient intake, malnutrition and communication problems. Weight loss, dehydration, mucosal ulceration, fluid-electrolyte imbalance may develop in patients who cannot be fed adequately, and total parenteral nutrition (TPN) can be started. Other important complications of oral mucositis are oral bleeding and infection. The ulcerated oral mucosa creates an entrance gate for microorganisms, increasing the risk of bacterial/fungal/viral infections. Infections may be limited only to the oral mucosa, as well as systemic infection and septicemia. As a result, the length of hospital stay of the patients increases, the treatment costs increase and their quality of life deteriorates. Therefore, early diagnosis of oral mucositis, planning and implementation of oral care are important. Responsibility of nurses in the management of oral mucositis; monitoring the oral cavity for symptoms, diagnosing mucositis, providing appropriate oral care, and educating patients.

In this context, it is extremely important to prevent oral mucositis, to evaluate the oral mucosa using a scale, and to reduce the degree of oral mucositis, that is, to perform appropriate oral care for its recovery, in terms of preventing other health problems and ensuring the well-being of the child. The aim of this thesis is to determine the effect of oral care with coconut oil on the degree of oral mucositis in pediatric oncology patients.

DETAILED DESCRIPTION:
Cancers have an important place among the childhood health problems. Although deaths in childhood cancers have decreased in recent years, it has been reported that the incidence of cancer has increased. Although the incidence of childhood cancers is lower than that of adult cancers, 0.5% of all cancer cases are children under the age of 15. Treatments such as chemotherapy, radiotherapy, surgical treatment, and bone marrow transplantation are applied alone or in combination in cancer treatment. Chemotherapy, which is one of the most used treatment methods in childhood cancers, destroys cancer cells, can prevent the spread of cancer cells in the body and the recurrence of the disease by 60-70%. Chemotherapy can cause complications by affecting normal cells and tissues as well as cancer cells. Among these complications, anemia, alopecia, dermatitis, thrombocytopenia, mucositis, nausea-vomiting and pain are the most common complications. Oral mucositis is one of the most common complications after chemotherapy and is seen in approximately 52% to 80% of children receiving treatment. Oral mucositis can directly affect the individual's quality of life by causing major problems such as shedding of the oral mucosal skin, ulceration, bleeding, pain, bacterial, fungal and viral infections in sick individuals. These problems make it difficult for the child to eat, drink, swallow and speak, and may lead to the development of biopsychosocial problems such as changes in comfort, decrease in body image and self-esteem, and increase in hospitalization time and hospital cost. It is important to prevent and manage mucositis in order to increase the quality of life of these children and reduce their stress levels. Proper oral hygiene and care practices are effective in the prevention and management of mucositis. Oral care provided by nurses is very important. Nurses, who play a primary role in patient care, are responsible for oral care and the prevention of mucositis. In order to prevent the development of mucositis, nurses need to have sufficient knowledge and skills, comply with practice protocols, take part in research that will form the basis of evidence, and follow the results of these studies. The aim of basic oral care is to reduce the effect of oral microbial flora and to prevent opportunistic infections. Basic oral care; It consists of brushing teeth with a soft-bristled toothbrush, cleaning between teeth with dental floss, rinsing the mouth using sterile water, saline or sodium bicarbonate. In basic oral care, it is recommended that the platelet (PLT) number be above 50,000 mm3 and the white blood cell (WBC) count over 1,000 mm3 for brushing and flossing. There is insufficient evidence that any component of basic oral care in the evidence-based practice guidelines fully prevents oral mucositis. However, there is evidence that it reduces the severity and duration of oral mucositis. To prevent and treat mucositis, saline, sodium bicarbonate, granulocyte colony stimulating factor (G-CSF), granulocyte-macrophage colony stimulating factor (GM-CSF), zinc sulfate, cryotherapy, sucralfate suspension, amifostine, prostaglandi E2 (PGE2) ), hydroxypropyl cellulose film, mucous sealants such as polyvinylpyrrolidone/sodium hyaluronate, topical application of vitamins A and E, parenteral application of β-carotene, low-dose laser therapy, glutamine, royal jelly, honey, aloe vera solution, omega-3 fatty acid, andiroba oil, black mulberry molasses and black mulberry syrup are used. In his study in 2020, Chadayan used coconut oil in his oral care to heal oral mucositis, and it was found that rinsing the mouth with coconut oil reduced the degree of oral mucositis. Studies have found that coconut oil has an effect on plaque formation and plaque-related gingivitis. Coconut oil is an edible oil and is consumed as part of the staple diet in many tropical countries. Coconut oil differs from most other dietary fats in that the predominant composition of coconut oil is a medium-chain fatty acid, while the basic building blocks of most other oils are almost entirely long-chain fatty acids. This is the physical and affect its chemical properties. Coconut oil contains 92% saturated acids, about 50% of which is lauric acid. Breast milk is the only other naturally occurring substance that contains such a high concentration of lauric acid. Lauric acid has proven anti-inflammatory effects and antimicrobial effects. These include Candida species and various viruses, including Helicobacter pylori, Staphylococcus aureus, Escherichia vulneris, Enterobcater and Candida glabrata, Candida albicans, Candida stellatoidea, Candida parapsilosis, Candida tropicalis, and Candida krusei. This study was planned to determine the effect of oral care with coconut oil on the degree of oral mucositis in pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between 7-18 years old,
* Having been diagnosed with cancer,
* Receiving chemotherapy at least every 21 or 28 days,
* Willingness and volunteering to participate in the study,
* Being able to speak Turkish and express himself

Exclusion Criteria:

* Not being healthy inside the mouth before chemotherapy,
* Being in terminal period,
* Being receiving radiotherapy
* Not willing or voluntarily to participate in the study,
* Not knowing Turkish.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
World Health Organization Oral Toxicity Scale | 21 day
  Evaluation of mucositis; It is performed by grading from 0 to 4 degrees according to the presence of erythema, ulceration, edema and pain. In the index, grade 0 indicates no mucositis, grade 1 mild, grade 2 moderate, grade 3-4 severe mucositis.
Children's International Mucositis Evaluation Scale (ChIMES) | 21 day
  1. The severity of intraoral pain; 2. The effect of pain on swallowing; 3. The effect of pain on eating; 4. The effect of pain on drinking; 5. The condition and reason for taking painkillers; 6. It consists of 6 items to evaluate the presence/absence of oral ulcers. Items 1, 2, 3 and 4 of ChIMES are each evaluated with a minimum of 0 and a maximum of 5 points; 5. Item is evaluated with a minimum of 0 and a maximum of 2 points; The 6th item is evaluated with the lowest 0 and the highest 1 point. When all items are answered, the minimum score from the scale is "0" and the maximum score is "23".

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ayçiçek, Prof. Dr., Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Cakmak S., Nural N. Oral Mucositis in Patients Receiving Chemotherapy and Radiotherapy: A Review. Dokuz Eylul University Faculty of Nursing Electronic Journal. 2020; 13(3): 185-194.
- [Background] Cavusoglu, H. Evidence-Based Nursing in the Management of Oral Mucositis. Turkiye Klinikleri Journal of Medical Sciences. 2007; 27(3): 398-406.
- [Background] Erdemir, F. and Taş Arslan, F. Pediatric Nursing: Child with Oncological Problems and Nursing Care. 2018; Ozyurt Publishing, Ankara
- [Background] Terracini B. Epidemiology of childhood cancer. Environ Health. 2011 Apr 5;10 Suppl 1(Suppl 1):S8. doi: 10.1186/1476-069X-10-S1-S8. PMID 21489218
- [Background] Türüner, E.K. and Büyükgönenç, L. Child Health Basic Nursing Approaches. Neyir Publishing. 2017; Ankara.
- [Background] Yavuz B, Bal Yilmaz H, Karaman N A study of reliability and validity for the Turkish version of children's international mucositisis evaluation scale for children with cancer. Turkish Journal of Oncology. 2011; 26(4): 157-162.
- [Result] Bayindir, S. The Effect of Oral Care with Black Mulberry Syrup on Oral Mucositis Healing in Individuals with COPD. Erciyes University, Institute of Health Sciences, Department of Nursing. 2018; PhD Thesis, Kayseri
- [Result] Albayrak, A. The effect of chewing gum with black mulberry syrup on the prevention of oral mucositis in children receiving chemotherapy. 2019; Unpublished master's thesis. Bursa Uludag University Institute of Health Sciences
- [Result] Baysal, E. The Effect of Cryotherapy on the Prevention of Oral Mucositis in Patients with Multiple Myeloma Diagnosed with Autologous Stem Cell Transplantation. Ege University Institute of Health Sciences, Department of Nursing Fundamentals. 2019; PhD Thesis, İzmir.
- [Result] Bektaş, M. The effect of planned basic oral care education given to children receiving chemotherapy on the prevention of oral mucositis. 2019; Master Thesis, Karadeniz Technical University, Institute of Health Sciences.
- [Result] Beşirik, S. & Canbulat Şahiner, N. Evidence-Based Practices in the Management of Mucositis in Children . Gumushane University Journal of Health Sciences. 2018; 7 (4), 128-133. Retrieved from https://dergipark.org.tr/tr/pub/gumussagbil/issue/41325/447904
- [Result] Chadayan, C. Effectiveness Of Coconut Oil Pulling On Oral Mucositis Among Cancer Patients In a Selected Hospital At Maduari.International Journal of Applied Research in Bioinformatics.2020. Doi:10.6084/m9.figshare.14769189.v1
- [Result] Devi KS, Allenidekania A. The Relationship of Oral Care Practice at Home with Mucositis Incidence in Children with Acute Lymphoblastic Leukemia. Compr Child Adolesc Nurs. 2019;42(sup1):56-64. doi: 10.1080/24694193.2019.1577926. PMID 31192726
- [Result] He M, Zhang B, Shen N, Wu N, Sun J. A systematic review and meta-analysis of the effect of low-level laser therapy (LLLT) on chemotherapy-induced oral mucositis in pediatric and young patients. Eur J Pediatr. 2018 Jan;177(1):7-17. doi: 10.1007/s00431-017-3043-4. Epub 2017 Nov 11. PMID 29128883
- [Result] Kobya Bulut H, Guducu Tufekci F. Honey prevents oral mocositis in children undergoing chemotherapy: A quasi-experimental study with a control group. Complement Ther Med. 2016 Dec;29:132-140. doi: 10.1016/j.ctim.2016.09.018. Epub 2016 Sep 19. PMID 27912937
- [Result] Kostak; M.A., Semerci; R., Eren T., Kocaaslan E.N. and Yıldız F. Effects of Oral Health Care Education on the Severity of Oral Mucositis in Pediatric Oncology Patients. 2020;Turkish Journal of Oncology. 35. 10.5505/tjo.2020.2366
- [Result] Mazhari F, Shirazi AS, Shabzendehdar M. Management of oral mucositis in pediatric patients receiving cancer therapy: A systematic review and meta-analysis. Pediatr Blood Cancer. 2019 Mar;66(3):e27403. doi: 10.1002/pbc.27403. Epub 2018 Nov 12. PMID 30421549
- [Result] Miller MM, Donald DV, Hagemann TM. Prevention and treatment of oral mucositis in children with cancer. J Pediatr Pharmacol Ther. 2012 Oct;17(4):340-50. doi: 10.5863/1551-6776-17.4.340. PMID 23413048
- [Result] Naseem M, Khiyani MF, Nauman H, Zafar MS, Shah AH, Khalil HS. Oil pulling and importance of traditional medicine in oral health maintenance. Int J Health Sci (Qassim). 2017 Sep-Oct;11(4):65-70. PMID 29085271
- [Result] Osmanoğlu Yurdakul, Z., Işık Esenay, F. Evidence-Based Methods Used for Oral Mucositis in Children with Cancer: A Systematic Review. Current Pediatrics. 2018; 16 (3), 51-78. Retrieved from https://dergipark.org.tr/tr/pub/pediatri/issue/40492/485516
- [Result] Peedikayil FC, Sreenivasan P, Narayanan A. Effect of coconut oil in plaque related gingivitis - A preliminary report. Niger Med J. 2015 Mar-Apr;56(2):143-7. doi: 10.4103/0300-1652.153406. PMID 25838632
- [Result] Ripari F, Filippone F, Zumbo G, Covello F, Zara F, Vozza I. The Role of Coconut Oil in Treating Patients Affected by Plaque-Induced Gingivitis: A Pilot Study. Eur J Dent. 2020 Oct;14(4):558-565. doi: 10.1055/s-0040-1714194. Epub 2020 Sep 22. PMID 32961569
- [Result] Shanbhag VK. Oil pulling for maintaining oral hygiene - A review. J Tradit Complement Med. 2016 Jun 6;7(1):106-109. doi: 10.1016/j.jtcme.2016.05.004. eCollection 2017 Jan. PMID 28053895
- [Result] Tomlinson D, Gibson F, Treister N, Baggott C, Judd P, Hendershot E, Maloney AM, Doyle J, Feldman B, Kwong K, Sung L. Refinement of the Children's International Mucositis Evaluation Scale (ChIMES): child and parent perspectives on understandability, content validity and acceptability. Eur J Oncol Nurs. 2010 Feb;14(1):29-41. doi: 10.1016/j.ejon.2009.10.004. Epub 2009 Dec 1. PMID 19955021
- [Result] Unal Çubukçu, N. & Çınar, S. Can oral mucositis be prevented in cancer patients receiving chemotherapy? . Clinical and Experimental Health Sciences. 2014; 2 (4), 155-163 . Retrieved from https://dergipark.org.tr/tr/pub/clinexphealthsci/issue/17851/187226
- [Result] Woolley J, Gibbons T, Patel K, Sacco R. The effect of oil pulling with coconut oil to improve dental hygiene and oral health: A systematic review. Heliyon. 2020 Aug 27;6(8):e04789. doi: 10.1016/j.heliyon.2020.e04789. eCollection 2020 Aug. PMID 32923724
- [Result] Yavuz B, Bal Yilmaz H. Investigation of the effects of planned mouth care education on the degree of oral mucositis in pediatric oncology patients. J Pediatr Oncol Nurs. 2015 Jan-Feb;32(1):47-56. doi: 10.1177/1043454214554011. Epub 2014 Nov 21. PMID 25416516